CLINICAL TRIAL: NCT07106320
Title: Evaluation of the Effect of Different Root Canal Irrigation Techniques on Periapical Tissue Healing and Postoperative Pain in Teeth With Apical Periodontitis
Brief Title: Evaluation of Different Root Canal Irrigation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, ASLI USTA TAHMAZ, Principal Investigator, Department of Endodontics, Medipol University, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-772.02-6497
Record Dates: First submitted 2025-07-12; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Apical Periodontitis
Keywords: Irrigation activation; Sonic activation; Ultrasonic activation; Apical periodontitis; Periapical Healing; Post operative pain
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasonic Irrigation Activation (VDW Ultra) (Experimental): Irrigation will be activated using an ultrasonic device (VDW Ultra) with an IRRI S tip positioned 2 mm short of the working length. Final irrigation protocol: Each canal receives a total of 6 mL of 3% Sodium Hypochlorite (NaOCl), will be delivered in three separate 2 mL portions. Each portion will be activated for 20 seconds. Subsequently, 2 mL of 17% Ethylenediaminetetraacetic Acid (EDTA) will be introduced into per canal and similarly activated ultrasonically for 20seconds to facilitate smear layer removal. As a final rinse, 5 mL of sterile saline will be used to flush out any residual irrigants and prevent potential chemical interactions.
  Interventions: Device: VDW Ultra Ultrasonic Irrigation Activation
- Sonic Irrigation Activation (EDDY) (Experimental): Irrigation will be activated using a sonic device (EDDY tip, VDW) positioned 2 mm short of the working length. Final irrigation protocol: Each canal receives a total of 6 mL of 3% Sodium Hypochlorite (NaOCl), will be delivered in three separate 2 mL portions. Each portion will be activated for 20 seconds. Subsequently, 2 mL of 17% Ethylenediaminetetraacetic Acid (EDTA) will be introduced into per canal and similarly activated for 20 seconds to facilitate smear layer removal. As a final rinse, 5 mL of sterile saline will be used to flush out any residual irrigants and prevent potential chemical interactions.
  Interventions: Device: EDDY Sonic Irrigation Activation
- Conventional Irrigation (Control) (Active Comparator): Irrigation will be performed using a syringe and needle without activation. Final irrigation will be performed using conventional syringe and needle irrigation without any activation. Each canal will be irrigated with 6 mL of 3% Sodium Hypochlorite (NaOCl), followed by 2 mL of 17% Ethylenediaminetetraacetic Acid (EDTA) and 5 mL of sterile saline, using a side-vented needle.
  Interventions: Procedure: Conventional Needle Irrigation

INTERVENTIONS:
Device: VDW Ultra Ultrasonic Irrigation Activation — Irrigation will be activated using an ultrasonic tip (IRRI S 21/25) connected to the VDW Ultra device (VDW GmbH, Munich, Germany), 2 mm short of working length. NaOCl and EDTA will each be activated for 20 seconds, repeated three times.
  Arms: Ultrasonic Irrigation Activation (VDW Ultra)
Device: EDDY Sonic Irrigation Activation — Irrigation solution will be activated using the EDDY sonic tip (VDW GmbH, Munich, Germany), positioned 2 mm short of the working length. NaOCl and EDTA will each be activated for 20 seconds, repeated three times.
  Arms: Sonic Irrigation Activation (EDDY)
Procedure: Conventional Needle Irrigation — Irrigation will be performed using a syringe and needle without activation. A total of 6 ml NaOCl, 2 ml EDTA and 5 mL of sterile saline will be used during final irrigation.
  Arms: Conventional Irrigation (Control)

SUMMARY:
This clinical study aims to evaluate the effect of different root canal irrigation techniques on postoperative pain levels and periapical healing in premolar and molar teeth diagnosed with apical periodontitis (Periapical Index (PAI) score 4-5). A total of 162 patients are randomly assigned to one of three groups: (1) sonic irrigation activation using EDDY, (2) ultrasonic irrigation activation using VDW Ultra, and (3) conventional syringe irrigation as the control. Postoperative pain will be recorded using the Visual Analog Scale (VAS) and Visual Analog Scale (VRS) at multiple time points up to one month. Periapical healing will be assessed using periapical imaging performed with the parallel technique one year after treatment. The study aims to determine whether enhanced irrigation techniques provide superior clinical outcomes compared to traditional methods.

DETAILED DESCRIPTION:
Root canal treatment aims to eliminate microorganisms and their byproducts from the complex root canal system to allow periapical tissue healing. Due to the anatomical complexity of root canals-such as isthmuses, apical deltas, and lateral canals-mechanical preparation alone is often insufficient. Therefore, chemical irrigation plays a vital role in successful disinfection.

This randomized clinical trial investigates the influence of three different irrigation protocols on postoperative pain and periapical healing in permanent premolar and molar teeth with radiographically evident apical periodontitis (Periapical Index (PAI) score 4-5).

The study includes three experimental groups :

Group 1 (Sonic activation): Irrigation solution is activated using the EDDY sonic tip.

Group 2 (Ultrasonic activation): Irrigation is activated using VDW Ultra ultrasonic tips.

Group 3 (Control): Conventional needle irrigation is performed without activation.

All treatments will be performed under rubber dam isolation and local anesthesia, using a standardized instrumentation protocol with ProTaper Next rotary files. Between each file change, the root canal will be irrigated with 5 ml of 3% sodium hypochlorite (NaOCl). The final irrigation protocol will be applied according to the assigned group. All endodontic procedures will be completed in a single session.

Postoperative pain levels will be assessed using both the Visual Analog Scale (VAS) and Visual Analog Scale (VRS) scales at 6, 12, 18, 24, 48, and 72 hours, as well as on day 7 and at 1 month. Patients will be asked to record analgesic consumption (400 mg ibuprofen as needed) and will submit pain diaries.

One year after treatment, periapical healing will be evaluated using periapical radiography (parallel technique) by two blinded observers.

.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Premolar and molar teeth with radiographically confirmed periapical lesions classified as Periapical Index (PAI) scores of 4 or 5 will be included in the analysis
* Systemically healthy individuals
* To be able to read and sign the informed consent form
* Physical and mental fitness to undergo treatment
* Willingness to attend all follow-up sessions

Exclusion Criteria:

* Patients with systemic diseases classified as ASA III or higher
* Presence of severe periodontal disease (probing depth >4 mm)
* Use of analgesics within the last 12 hours or antibiotics within the past month before the treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Periapical Healing | From end of treatment to 1 year
  The primary outcome of this study is periapical healing. It will be assessed radiographically using standardized periapical images (taken with the parallel technique), captured preoperatively and at the 1-year follow-up, and evaluated using the Periapical Index (PAI) score by two blinded observers. The PAI score ranges from 1 (healthy periapical structures) to 5 (severe periodontitis).

SECONDARY OUTCOMES:
Postoperative Pain Intensity - Visual Analog Scale | From end of treatment to 6, 12, 18, 24, 48, and 72 hours; 7 days; and 1 month after root canal treatment
  The secondary outcome is postoperative pain intensity. Pain will be assessed at multiple time points (6, 12, 18, 24, 48, and 72 hours, and at 1 week and 1 month post-treatment) using Visual Analog Scale (VAS) where 0 represents "no pain" and 10 represents "worst imaginable pain".

OTHER OUTCOMES:
Post Operative Pain İntensity | From end of treatment to 6, 12, 18, 24, 48, and 72 hours; 7 days; and 1 month after root canal treatment
  The secondary outcome is postoperative pain intensity. Pain will be assessed at multiple time points (6, 12, 18, 24, 48, and 72 hours, and at 1 week and 1 month post-treatment) using Verbal Rating Scale (VRS), which categorizes pain into four levels: 0 (no pain), 1 (mild), 2 (moderate), and 3 (severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD), including all IPD that underlie the results reported in the publication
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared starting 6 months after publication.
Access Criteria: Qualified researchers may request access to all de-identified individual participant data (IPD) and study protocols. Access will be granted upon reasonable request by contacting the corresponding author via email and after signing a data sharing agreement